CLINICAL TRIAL: NCT04373694
Title: Pain Perception During Vaginoscopy Compared to Traditional Hysteroscopy for Hysteroscopy Morcellation in Outpatient Clinic: A Randomized Trial
Brief Title: Vaginoscopy Compared to Traditional Hysteroscopy for Hysteroscopy Morcellation in Outpatient Clinic. A Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.380
Record Dates: First submitted 2020-04-23; First posted 2020-05-04 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Leiomyoma of Uterus
Keywords: vaginoscopy; hysteroscopy morcellation; infertile population
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard hysteroscopy (Active Comparator): morcellation hysteroscopy with intravenous sedation and paracervical bloc
  Interventions: Procedure: standard hysteroscopy
- Vaginoscopy (Experimental): morcellation hysteroscopy with only intravenous sedation
  Interventions: Procedure: vaginoscopy

INTERVENTIONS:
Procedure: vaginoscopy — vaginal distension with hysteroscope for hysteroscopy morcellation (without speculum or tenaculum forceps)
  Arms: Vaginoscopy
Procedure: standard hysteroscopy — speculum, paracervical block before hysteroscopy morcellation
  Arms: Standard hysteroscopy

SUMMARY:
This study is a randomized controlled trial take place in a fertility outpatient clinic in an academic hospital. Women between 18 and 52 years old requiring polypectomy or myomectomy by hysteroscopy morcellation for abnormal uterine bleeding or for fertility issue are included. The aim is to evaluate pain perception between vaginal and traditional hysteroscopy for hysteroscopic morcellation. The investigator's hypothesis is that pain perception is lower using vaginoscopy compared to traditional hysteroscopy.

DETAILED DESCRIPTION:
78 participants will be randomised in two groups:

1. traditional hysteroscopy: under intravenous sedation, hysteroscopic morcellation is perform after speculum insertion, vaginal cleansing, and paracervical anesthesia with xylocain 1%.
2. Vaginal hysteroscopy: under intravenous sedation, hysteroscopic morcellation is perform after vaginal cleansing using vaginal distension with saline solution

In addition to pain perception, other outcomes includes: complication rates, time to continue fertility treatment, time to pregnancy

ELIGIBILITY:
Inclusion Criteria:

* polyp or fibroid previously diagnosed by hysteroscopy
* polyp less than 2 cm
* submucosal fibroid (type 0 or 1 according to the 2011 FIGO uterine fibroid classification) less than 2 cm
* if more than 1 fibroid: total fibroid have to be less or equal 4 cm

Exclusion Criteria:

* cervical stenosis
* polyp or fibroid more than 2 cm
* pregnancy
* blood dyscrasia

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in pain perception between vaginoscopy group and traditional hysteroscopy group | immediately after intervention
  10 point visual analog pain scale: 0 for no pain to 10 for unbearable pain

SECONDARY OUTCOMES:
Difference in length of time of procedure between vaginoscopy group and traditional hysteroscopy group | immediately after intervention
  length of time in minutes between start and end of procedure including morcellation
Difference in proportion of vasovagal syncope between vaginoscopy group and traditional hysteroscopy group | immediately after surgery
  Presence of jerky abnormal movements or a slow weak pulse rate associated to at least one symptoms: nausea, pale skin, blurred vision, warm feeling or cold sweat.
Difference in proportion of uterine perforation between vaginoscopy group and traditional hysteroscopy group | immediatly after surgery
  presence of one or more signs during intervention: extension of the instrument goes beyong the limitation of the uterus, loss of resistance, sudden loss of vision, direct visualisation of the perforation
Difference in length of time to continue fertility treatment between vaginoscopy group and traditional hysteroscopy group | up to 1 year
  length of time in months to continue fertility treatment after procedure
Difference in length of time to pregnancy between vaginoscopy group and traditional hysteroscopy group | up to 1 year
  length of time in months to be pregnant after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carole KAMGA-NGANDE, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- CHUM - Clinique Médecine et biologie de la reproduction, Montreal, Quebec, Canada